CLINICAL TRIAL: NCT03644017
Title: Prospective Investigation of The Merit WRAPSODY™ Endovascular Stent Graft for Treatment of Venous Outflow Circuit Obstruction In Hemodialysis Patients
Brief Title: The Merit WRAPSODY™ Endovascular Stent Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merit Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVO-P1-18-01
Record Dates: First submitted 2018-08-16; First posted 2018-08-23 (Actual); Results first posted 2021-07-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2021-12

CONDITIONS: Venous Stenosis; Venous Occlusion
Keywords: Dialysis; Venous Stenosis; Venous Occlusion; Stent Graft

STUDY DESIGN:
Intervention Model Description: Single arm treated with investigational device WRAPSODY Stent Graft
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- WRAPSODY Stent Graft (Experimental): All subjects will receive treatment via WRAPSODY Stent Graft Placement.
  Interventions: Device: WRAPSODY Stent Graft Placement

INTERVENTIONS:
Device: WRAPSODY Stent Graft Placement — The stent graft will be placed into a target lesion (stenosis or occlusion) of a vein
  Other Names: Stent Graft; Covered Stent

SUMMARY:
This is a phase 1 study, designed to evaluate the safety and effectiveness of the WRAPSODY Stent Graft for the treatment of venous outflow circuit obstructions in the veins of the arm or thoracic central veins of subjects who receive chronic dialysis treatment for end stage renal disease.

DETAILED DESCRIPTION:
The study will consist of a screening period in which subject eligibility will be determined. Approximately 50 subjects meeting the study entry criteria will be enrolled. Placement of the WRAPSODY stent graft will follow the procedure. Post study procedure subjects will have planned follow-up visits at 30 days, 3, 6 and 12months, and additional visits as referred by the subject's dialysis facility.

The primary study safety endpoint will be the proportion of subjects without any localized or systemic safety events through 30 days that affect the access or venous outflow circuit and resulted in surgery, hospitalization, or death. Subjects will continue to be followed up to 12 months for supplementary information.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has signed informed consent
2. Subject is ≥ 21 years of age
3. Subject is undergoing chronic hemodialysis or other forms of renal replacement therapy including transplantation and has one of the following being used: a. AV graft placed in the arm ≥30 days prior OR b. Mature fistula in the arm with at least one successful dialysis session completed
4. Angiographic evidence of stenosis
5. The target lesion has ≥ 50% stenosis
6. Subject has clinical or hemodynamic evidence of a venous outflow stenosis or obstruction
7. Full expansion of an appropriately sized standard angioplasty balloon has been achieved during primary angioplasty at the target lesion prior to enrollment

Exclusion Criteria:

1. Subject has undergone an intervention (surgical or percutaneous) of the AVF/AVG <30 days from the date of the initial study procedure
2. Subject has had a previous stent or stent graft placed in the venous outflow circuit ≤30 days from the date of the initial study procedure
3. Active hemodialysis access is not in the arm
4. A pseudoaneurysm is present within the target lesion
5. Target lesion is in SVC, IJV, under the clavicle, across the elbow, in the needling segment of AVF or AVG anastomosis, located within a stent
6. Lesions, other than the target lesion, in the venous outflow circuit with >30% stenosis
7. Known or suspected infection of the hemodialysis access site and/or septicemia
8. Permanent pacemaker or automated implantable cardioverter defibrillator (AICD) on the side with the target lesion
9. Current central venous catheter for dialysis access
10. Uncorrectable coagulation disorders
11. Hypersensitivity to nickel titanium alloy
12. The subject is enrolled in another investigational study
13. The subject is unable or unwilling to comply with the protocol requirements
14. Life expectancy is ≤ 12 months
15. Subject cannot receive heparin or equivalent anticoagulant
16. Allergy to radiographic contrast material which cannot be adequately premedicated
17. Subject is pregnant, breastfeeding, or pre-menopausal and intending to become pregnant
18. Subject's access is anticipated to be abandoned within 3 months
19. Subject has a thoracic central vein obstruction that would lead to stent graft placement across the internal jugular vein
20. Subject's hemodialysis access is thrombosed
21. Active malignancy other than non-melanomatous skin cancer
22. Any other condition deemed exclusionary in the opinion of the investigator

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2021-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James A Gilbert, MD, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (3):
- G. Gennimatas General Hospital of Athens, Athens, Greece
- United Kingdom (2):
  - Queen Elizabeth University Hospital, Glasgow
  - Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | WRAPSODY Stent Graft
Started | 46
Completed | 39
Not Completed | 7
Not completed — Access Abandonment | 5
Not completed — Kidney Transplant | 2

BASELINE CHARACTERISTICS:
Arm/Group | WRAPSODY Stent Graft
Number analyzed (Participants) | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.7 (12.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 45
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 39
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Greece | 23
  United Kingdom | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Without Any Localized or Systemic Safety Events Through 30 Days
Description: The total number of subjects without any localized or systemic safety events through 30 days that affect the access or venous outflow circuit and resulted in surgery, hospitalization, or death
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | WRAPSODY Stent Graft
Number analyzed (Participants) | 46
Participants | 45

2. Primary Outcome: Number of Participants With Target Lesion Primary Patency at 30 Days
Description: The total number of subjects with Target Lesion Primary Patency at 30 days
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | WRAPSODY Stent Graft
Number analyzed (Participants) | 45
Participants | 45

3. Secondary Outcome: Number of Participants With Target Lesion Primary Patency at 3 Months
Description: The total number of subjects with Target Lesion Primary Patency at 3 months
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | WRAPSODY Stent Graft
Number analyzed (Participants) | 44
Participants | 44

4. Secondary Outcome: Number of Participants With Target Lesion Primary Patency at 6 Months
Description: The total number of subjects with Target Lesion Primary Patency at 6 months
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | WRAPSODY Stent Graft
Number analyzed (Participants) | 43
Participants | 42

5. Secondary Outcome: Number of Participants With Target Lesion Primary Patency at 12 Months
Description: The total number of subjects with Target Lesion Primary Patency at 12 months
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | WRAPSODY Stent Graft
Number analyzed (Participants) | 39
Participants | 33

6. Secondary Outcome: Number of Participants With Assisted Target Lesion Primary Patency at 30 Days
Description: The total number of subjects with Assisted Primary Patency of the Target Lesion at 30 days
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | WRAPSODY Stent Graft
Number analyzed (Participants) | 45
Participants | 45

7. Secondary Outcome: Number of Participants With Assisted Target Lesion Primary Patency at 3 Months
Description: The total number of subjects with Assisted Primary Patency of the Target Lesion at 3 months
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | WRAPSODY Stent Graft
Number analyzed (Participants) | 44
Participants | 44

8. Secondary Outcome: Number of Participants With Assisted Target Lesion Primary Patency at 6 Months
Description: The total number of subjects with Assisted Primary Patency of the Target Lesion at 6 months
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | WRAPSODY Stent Graft
Number analyzed (Participants) | 43
Participants | 43

9. Secondary Outcome: Number of Participants With Assisted Target Lesion Primary Patency at 12 Months
Description: The total number of subjects with Assisted Primary Patency of the Target Lesion at 12 months
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | WRAPSODY Stent Graft
Number analyzed (Participants) | 39
Participants | 39

10. Secondary Outcome: Number of Participants With Access Circuit Primary Patency at 30 Days
Description: The total number of subjects with Access Circuit Primary Patency at 30 days
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | WRAPSODY Stent Graft
Number analyzed (Participants) | 45
Participants | 43

11. Secondary Outcome: Number of Participants With Access Circuit Primary Patency at 3 Months
Description: The total number of subjects with Access Circuit Primary Patency at 3 months
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | WRAPSODY Stent Graft
Number analyzed (Participants) | 45
Participants | 40

12. Secondary Outcome: Number of Participants With Access Circuit Primary Patency at 6 Months
Description: The total number of subjects with Access Circuit Primary Patency at 6 months
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | WRAPSODY Stent Graft
Number analyzed (Participants) | 45
Participants | 38

13. Secondary Outcome: Number of Participants With Access Circuit Primary Patency at 12 Months
Description: The total number of subjects with Access Circuit Primary Patency at 12 months
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | WRAPSODY Stent Graft
Number analyzed (Participants) | 44
Participants | 29

14. Secondary Outcome: Number of Participants With Assisted Access Circuit Primary Patency at 30 Days
Description: The total number of subjects with Assisted Access Circuit Primary Patency at 30 days
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | WRAPSODY Stent Graft
Number analyzed (Participants) | 45
Participants | 45

15. Secondary Outcome: Number of Participants With Assisted Access Circuit Primary Patency at 3 Months
Description: The total number of subjects with Assisted Access Circuit Primary Patency at 3 months
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | WRAPSODY Stent Graft
Number analyzed (Participants) | 45
Participants | 44

16. Secondary Outcome: Number of Participants With Assisted Access Circuit Primary Patency at 6 Months
Description: The total number of subjects with Assisted Access Circuit Primary Patency at 6 months
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | WRAPSODY Stent Graft
Number analyzed (Participants) | 45
Participants | 43

17. Secondary Outcome: Number of Participants With Assisted Access Circuit Primary Patency at 12 Months
Description: The total number of subjects with Assisted Access Circuit Primary Patency at 12 months
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | WRAPSODY Stent Graft
Number analyzed (Participants) | 44
Participants | 39

18. Secondary Outcome: Number of Participants With Clinical Success
Description: The resumption of successful dialysis through existing access for at least one session following the initial study procedure
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | WRAPSODY Stent Graft
Number analyzed (Participants) | 45
Participants | 45

19. Secondary Outcome: Number of Participants With Anatomic Success
Description: Less than 30% residual stenosis immediately following the study procedure
Time Frame: Immediately following the study procedure
Measure: Count of Participants; unit: Participants
Arm/Group | WRAPSODY Stent Graft
Number analyzed (Participants) | 46
Participants | 46

20. Secondary Outcome: Number of Participants With Procedural Success
Description: The achievement of both clinical and anatomic success
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | WRAPSODY Stent Graft
Number analyzed (Participants) | 45
Participants | 45

21. Other Pre Specified Outcome: Number of Participants With Stent Graft Integrity (Subset of Subjects With Thoracic Central Venous Target Lesions Only)
Description: Total number of participants (subset of subjects with thoracic central venous target lesions only) with freedom from stent graft fracture, defined as clear interruption of a stent strut observed in a minimum of two projections taken during the 12 month visit or after determined by DMC/CEC examination of X-Ray images.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | WRAPSODY Stent Graft
Number analyzed (Participants) | 8
Participants | 8

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | WRAPSODY Stent Graft
All-Cause Mortality (participants affected / at risk) | 0/46
Serious Adverse Events (participants affected / at risk) | 10/46
Other Adverse Events (participants affected / at risk) | 0/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WRAPSODY Stent Graft (N=46)
Pneumonia (Infections and infestations) | 3 (3)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Myocardial infarction (Cardiac disorders) | 1 (1)
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 2 (2)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Device dislocation (Product Issues) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Coronavirus test positive (Investigations) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-07): https://cdn.clinicaltrials.gov/large-docs/17/NCT03644017/Prot_SAP_000.pdf